CLINICAL TRIAL: NCT03707106
Title: An Efficacy Study Using an Established Cognitive Behavioral Therapy Manual for Smoking Cessation Comparing the Benefit of Virtual Reality Cue Exposure to a Specific Stress Reduction Protocol for Relapse Prevention
Brief Title: Benefits of a Cognitive Behavioral Therapy Intervention for Smoking Cessation Supported by Virtual Reality Smoking Cue Exposure
Acronym: ViReTa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University of Regensburg (Other)
Responsible Party: Principal Investigator, Anil Batra, Deputy Head of Psychiatry, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 70111871
Record Dates: First submitted 2018-04-05; First posted 2018-10-16 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Smoking Cessation
Keywords: virtual reality; cue exposure; progressive muscle relaxation
MeSH Terms: conditions — Smoking Cessation | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR based cue exposure smoking cessation (Experimental): an established CBT intervention for smoking cessation supported by cue exposure in virtual reality
  Interventions: Behavioral: CBT smoking cessation; Behavioral: virtual reality based cue exposure
- PMR supported smoking cessation (Active Comparator): an established CBT intervention for smoking cessation supported supported by specific stress reduction (Progressive Muscle Relaxation, Jacobson)
  Interventions: Behavioral: CBT smoking cessation; Behavioral: progressive muscle relaxation

INTERVENTIONS:
Behavioral: CBT smoking cessation — an established protocol for smoking cessation based on cognitive behavioral therapy
Behavioral: virtual reality based cue exposure — smoking cue exposure in virtual reality
  Arms: VR based cue exposure smoking cessation
Behavioral: progressive muscle relaxation — Progressive muscle relaxation for unspecific stress reduction
  Arms: PMR supported smoking cessation

SUMMARY:
Cognitive-behavioral therapy (CBT) combined with medication is an established intervention for smoking cessation. However, long-term abstinence rates of maximum 35% are yielded. Moreover, acceptance of drug treatment is partly very low. Professional recommendation of drug treatment besides nicotine-replacement aids is restrained considering side effects and contraindications. Currently, cue exposure is highly discussed as intervention for craving reduction supporting CBT. There is evidence for benefits of cue exposure optimizing smoking cessation outcomes, as well as evidence for efficacy of exposure in virtual reality (VR) up to date.

However, this is the first randomized controlled study focusing on efficacy increases by VR cue exposure supporting an established CBT smoking cessation manual. The control group receives a specific stress reduction treatment (independent of smoking cues), namely, the Progressive Muscle Relaxation (PMR, according to Jacobson) additionally to the established smoking cessation CBT.

ELIGIBILITY:
Inclusion Criteria:

* daily smokers for at least 2 years, smoking minimum 10 cigarettes a day

Exclusion Criteria:

* pregnancy
* current participation in another smoking cessation program within 6 months before assignment
* current diagnosis of a psychiatric disease including a depression or substance use disorder (excluding nicotine dependency)
* lifetime diagnosis of a psychiatric disease : psychosis, bipolar affective disorder, posttraumatic stress disorder, conversion disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Continuous (self-reported) abstinence rates from smoking 6 months after end of treatment | at the 6 month follow-up
  6-month continuous smoking abstinence according to the Russell Standard (West et al., 2005): no cigarette smoking assessed by self-report (number of smoked cigarettes) and a negative biochemical validation (CO measurement below 9) at the ﬁnal follow-up. 6-month continuous smoking abstinence ordinal scale: 0=no abstinence, 1= either subjective or biochemical validation depicts no abstinence, 2= biochemical validated abstinence at the 6 months follow-up.

SECONDARY OUTCOMES:
Changes in smoking cue event-related potentials (ERP: LPP) | Differences from baseline to the 6 month follow-up
  late positive potential (LPP) amplitude (Microvolts)
Changes in smoking cue event-related potentials (ERP:P3) | Differences from baseline to the 6 month follow-up
  P3 amplitude (Microvolts) during avoidance of smoking cues
Changes in approach tendency to smoking pictures | Differences from baseline to the 6 month follow-up
  Difference in reaction time (ms) bias berween neutral and smoking condition. Approach Bias is calculated as reaction time (ms) difference in avoidance and approach condition.
Changes in smoking cue reactivity related skin conductance level | Differences from baseline to the 6 month follow-up
  Differences in conductance level (MicroSiemens) during smoking cue exposure and exposure to a neutral cue.
Changes in Theta and Alpha band power during smoking cue exposure | Differences from baseline to the 6 month follow-up
  Differences in Alpha and Theta band power during smoking cue exposure and neutral cue exposure.
Changes in heartbeat-evoked potential during smoking cue exposure | Differences from baseline to the 6 month follow-up
  Amplitude (microvolts) of heartbeat-evoked potential
Subjective ratings on the smoking self-efficacy scale | Differences from baseline to the 6 month follow-up
  Subjective ratings on on the German version of the self-efficacy scale for smoking cessation (Jäkle et al., 1999) total score for the questionnaire: minium total score (sum): 9 (low self-efficacy, worse outcome), maximum total score= 45 (high self-efficacy, better outcome)
Number of daily smoked cigarettes after smoking cessation | Time Frame: Differences from smoking cessation to the 6 month follow-up
  Sum of self-reported smoked cigarettes after smoking cessation

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - University Regensburg, Regensburg

REFERENCES:
- [Derived] Kroczek AM, Schroder B, Rosenbaum D, Muhleck A, Diemer J, Muhlberger A, Ehlis AC, Batra A. Virtual reality cue exposure as an add-on to smoking cessation group therapy: a randomized controlled trial. Addict Sci Clin Pract. 2025 Apr 11;20(1):34. doi: 10.1186/s13722-025-00561-2. PMID 40211338